CLINICAL TRIAL: NCT02418832
Title: Rete Testis Needle Aspiration for Retrieval of Sperm in Men With Azoospermia Using Ultrasound Guidance
Brief Title: Testis Needle Aspiration of Sperm in Men With Azoospermia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Benjamin Reubinoff, Professor, Chairman of the Department of Obstetrics and Gynecology, Hadassah Ein Kerem, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0238-13-HMO
Record Dates: First submitted 2015-03-12; First posted 2015-04-16 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Azoospermia
Keywords: Azoospermia; Rete Testis; TEFNA
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with Azoospermia, sperm cell aspiration and TEFNA (Other): Men between 16-80 with Obstructive and Non-Obstructive Azoospermia; Sperm cell aspiration,TEFNA and Ultrasound Guidance
  Interventions: Procedure: Sperm cell aspiration and TEFNA

INTERVENTIONS:
Procedure: Sperm cell aspiration and TEFNA — Testicular Fine Needle Aspiration (TEFNA)

SUMMARY:
Needle aspiration of the epididymis causes rupture and irreversible damage to the duct. Recurring punctures and needle aspirations of fluid and tissue during Testicular Fine Needle Aspiration (TEFNA) procedure cause irreparable injury and loss of part of the testis' tubules. The hypothesis of this research is that production of sperm from the testis will be improved due to ultrasonically guided Rete Testis needle aspiration. In cases of Obstructive Azoospermia, the Rete Testis is expected to contain a large number of sperm cells. In cases of Non-Obstructive Azoospermia, the investigators can expect to produce sperm cells from aspiration of the Rete Testis, which drains all of the testis' tubules. Furthermore, catheterization of the Rete Testis will allow for the drainage of all testes tubules and for the production of sperm cells created locally in some of the tubules or in parts of them.

The potential advantage of needle aspiration from the Rete Testis is that the procedure will allow for the aspiration from all the testes tubules, as opposed to the standard method of sperm cells production from the testis which samples only some of the tubules. Therefore, it is expected that the procedure suggested in this research will be more efficient than the standard procedures currently in practice. An additional advantage to this procedure is that puncture and aspiration of the tubule network is not expected to block the drainage from the testis, as is the case in aspiration of the epididymis, and it is also not expected to damage the tubules, as is the case in TEFNA and in TESE.

DETAILED DESCRIPTION:
Potential subjects will be Azoospermic men who turn to the IVF unit at Hadassah Ein Kerem and are candidates for a TEFNA treatment.

Only after the men will receive an explanation of the TEFNA procedure and sign a consent form for TEFNA will they be invited to join the study.

After an explanation, the men will sign a consent form (attached) for participation in the study.

The TEFNA procedure in each testis will begin with an ultrasonically guided Rete Testis needle aspiration and washing of the testes tubules. A PP Spinal Needle, of 20-27 Gage and 90mm length, will be used for the ultrasonically guided puncture of the testis and catheterization of the Rete Testis network. After the catheterization, there will be an aspiration, followed by the washing of the testis tubule network in saline used for IV, in a volume of up to 1mL (5), using a 1mL syringe. In men with Obstructive Azoospermia, in case the samples aspirated from the Rete Testis will contain many motile sperm cells (more than hundreds), there will be no need for a TEFNA procedure. In cases where an initial sample of the Rete Testis aspiration will not show many motile sperm cells, the TEFNA procedure will continue on as planned.

The samples from the Rete Testis aspiration will be separately checked for sperm cells from the sample and tissue produced from the TEFNA procedure. The sperm cells produced from the Rete Testis will be used for cryopreservation or fertilization of the ovum of the patient's partner, as is customary in sperm cells attained through the TEFNA procedure. Should sperm cells be produced both from the Rete Testis and from the epididymis or testes, the partner's ovum will be fertilized by the highest quality sperm cells of both sources.

Clinical follow-up on patients will be conducted as customary after testis aspiration.

The patients will be invited six months after the procedure for an ultrasonic check-up of the testes and the Rete Testis.

ELIGIBILITY:
Inclusion Criteria:

* Men with Obstructive/Non-Obstructive Azoospermia who turned to sperm cell aspiration for IVF and were found suitable for TEFNA and signed consent form.

Exclusion Criteria:

* healthy, non-azoospermic men
* men who are unsuitable for the TEFNA procedure
* men who don't sign the Informed Consent

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-07-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Guidance of Sperm Aspiration to Improve Efficiency of TEFNA | 5 years
  The efficiency will be assessed by the percentage of participants in which at least one sperm cell will be successfully retrieved from ultrasound-guided Rete-Testis aspiration. The efficiency will be calculated separately for participants with Obstructive- and non-Obstructive Azoospermia.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E. Reubinoff, MD PhD, Principal Investigator — Hadassah University Medical Center
Locations (1):
- Hadassah University Medical Center, Ein Kerem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoysman R, Van Roosendaal E, Bollen N, Vandervorst M, Vanderzwalmen P, Standaert V, Berting G, Debauche C, Lefere C. Modern sperm retrieval techniques and their usefulness in oocyte fertilization. BJU Int. 2001 Jul;88(2):141-6. doi: 10.1046/j.1464-410x.2001.02301.x. No abstract available. PMID 11446872
- [Background] Lewin A, Reubinoff B, Porat-Katz A, Weiss D, Eisenberg V, Arbel R, Bar-el H, Safran A. Testicular fine needle aspiration: the alternative method for sperm retrieval in non-obstructive azoospermia. Hum Reprod. 1999 Jul;14(7):1785-90. doi: 10.1093/humrep/14.7.1785. PMID 10402390
- [Background] Friedler S, Raziel A, Strassburger D, Soffer Y, Komarovsky D, Ron-El R. Testicular sperm retrieval by percutaneous fine needle sperm aspiration compared with testicular sperm extraction by open biopsy in men with non-obstructive azoospermia. Hum Reprod. 1997 Jul;12(7):1488-93. doi: 10.1093/humrep/12.7.1488. PMID 9262283
- [Background] Schlatt S, Rosiepen G, Weinbauer GF, Rolf C, Brook PF, Nieschlag E. Germ cell transfer into rat, bovine, monkey and human testes. Hum Reprod. 1999 Jan;14(1):144-50. doi: 10.1093/humrep/14.1.144. PMID 10374111
- [Background] Hermann BP, Sukhwani M, Winkler F, Pascarella JN, Peters KA, Sheng Y, Valli H, Rodriguez M, Ezzelarab M, Dargo G, Peterson K, Masterson K, Ramsey C, Ward T, Lienesch M, Volk A, Cooper DK, Thomson AW, Kiss JE, Penedo MC, Schatten GP, Mitalipov S, Orwig KE. Spermatogonial stem cell transplantation into rhesus testes regenerates spermatogenesis producing functional sperm. Cell Stem Cell. 2012 Nov 2;11(5):715-26. doi: 10.1016/j.stem.2012.07.017. PMID 23122294